CLINICAL TRIAL: NCT02659163
Title: An Integrated Closed-loop Feedback System for Pediatric Cardiometabolic Disease
Acronym: STRIVE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Nicolas M. Oreskovic, MD, MPH, Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HS024001 (AHRQ)
Record Dates: First submitted 2016-01-12; First posted 2016-01-20 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Health Behavior
Keywords: cardiometabolic risk; obesity; mHealth; health behaviors
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Intervention subjects will receive feedback on their health behaviors along with clinical recommendations.
  Interventions: Behavioral: mHealth wristband; Behavioral: mHealth scale; Behavioral: EMA; Behavioral: mHealth app; Behavioral: Integrated closed-loop feedback system
- control (Active Comparator): Control subjects will receive feedback on their health behaviors for self-guided care.
  Interventions: Behavioral: mHealth wristband; Behavioral: mHealth scale; Behavioral: EMA; Behavioral: mHealth app; Behavioral: Health Behavior Feedback

INTERVENTIONS:
Behavioral: mHealth wristband — A wristband containing several sensors worn by participants to collect daily objective patient-generated health behavior data on physical activity, sleep, and screen time
  Other Names: sensors
Behavioral: mHealth scale — A wireless scale used by participants to measure and record daily weight.
  Other Names: wireless sscale
Behavioral: EMA — Self-reported information on sugar sweetened beverage consumption collected via mobile messaging
  Other Names: Sugar Sweetened Beverage Assessment
Behavioral: mHealth app — A mobile application that houses study data and provides two-way messaging between the study team and study participants.
Behavioral: Health Behavior Feedback — Provide feedback on patient-generated health behaviors data, along with standard of care recommendations, for self-guided
  Arms: control
Behavioral: Integrated closed-loop feedback system — Daily feedback and weekly e-report cards on patient-generated longitudinal health behaviors along with clinical recommendations via mobile messaging
  Arms: intervention

SUMMARY:
The high prevalence and burden of cardiometabolic disease underlie the urgent need to identify novel approaches to managing and preventing cardiometabolic disease and risk. This project will test an innovative use of mobile health technology to implement a closed-loop feedback system that collects objective patient-generated data and provides clinical recommendations to modify contributing health behaviors. In addition to improving care for cardiometabolic disease, the tools and methods developed by this study for collecting patient data and providing clinical feedback could also easily be adapted and applied to a range of other health conditions, and are thus highly relevant to public health.

DETAILED DESCRIPTION:
Cardiometabolic disease - a clustering of medical conditions and risk factors which includes obesity, diabetes, impaired liver function, and an increased risk in children for adult-onset cardiovascular disease - represents a major population-wide health burden in the United States. Management of cardiometabolic disease also imposes a substantial financial burden on the economy and ties up significant healthcare resources. It is well-known that many of the lifestyle and health behaviors that contribute to cardiometabolic disease are difficult to modify once established, and childhood represents an opportune time for promoting healthy behaviors. Patient-centered outcomes research (PCOR) has identified certain health behaviors as important and actionable in modifying cardiometabolic risk, namely weight management, physical activity, screen-time, sleep, and consumption of sugar-sweetened beverages. Mobile health technology (mHealth) could be used to monitor and counsel on common health behaviors associated with cardiometabolic risk, which may facilitate the inclusion of PCOR evidence on cardiometabolic disease into clinical practice. The overall goal of this research is to use mHealth technology to accelerate the uptake of PCOR findings on treatment of cardiometabolic disease. To achieve our goal, this study will develop a novel set of mHealth tools capable of collecting health behavior information and determine to what extent providing clinical feedback on these health behaviors improves obesity and health behaviors among children ages 6-12 year and their families. In this study we will develop, implement, and test the comparative clinical effectiveness of a closed-loop feedback system for collecting patient data and providing recommendations. The specific aims of this study are: 1) to develop an integrated closed-loop feedback system that incorporates longitudinal mHealth data in managing cardiometabolic disease among at-risk families, and 2) to determine the extent to which an integrated closed-loop system that provides feedback on objective patient-generated data improves cardiometabolic risk, as measured by changes in body mass index and health behaviors including, physical activity, screen-time, sleep, and sugar-sweetened beverage consumption. This research will develop novel mHealth tools and approaches that will allow healthcare providers and patients to better understand disease risk and improve disease management by collecting patient data 1) repeatedly over time, 2) simultaneously, and 3) objectively. This study is innovative because it will use mHealth tools to simultaneously collect longitudinal data on multiple health behaviors known to be associated with cardiometabolic risk, and it will offer a new approach to implementing and disseminating PCOR findings via a novel closed-loop feedback system. The high prevalence of cardiometabolic disease makes this innovative closed-loop system very relevant to public health. The mHealth tools and methods developed by this study for collecting patient data and providing clinical feedback could also easily be adapted and applied to a range of other health conditions.

ELIGIBILITY:
Inclusion Criteria:

* ages 6-12 years
* body mass index categorized as overweight or obese
* followed for obesity care
* an adult household family member with one or more elevated cardiometabolic risk, as defined by established or documented increased risk of cardiometabolic disease (overweight, obesity, hypertension, coronary artery disease, diabetes or glucose intolerance, dyslipidemia, non-alcoholic fatty liver disease, cerebrovascular disease)
* participating parent must own Android Smartphone
* Wi-Fi access at home
* speak and read English

Exclusion Criteria:

* n/a

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
BMI, Child | 6 months
  mean change in BMI z-score

SECONDARY OUTCOMES:
Health Behaviors Index, Child and Adult | 6 months
  Cardiometabolic risk will be reported as an index score, a continuous variable calculated as the sum of Z-scores of mean daily moderate-to-vigorous physical activity (minutes), mean daily sleep (minutes), mean daily screen time (minutes), and mean weekly sugar sweetened beverage intake.
BMI, Adult | 6 months
  mean change in BMI z-score

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Oreskovic, MD, MPH, Principal Investigator — Massachusetts General Hospital